CLINICAL TRIAL: NCT06093178
Title: Assessing the Feasibility of a Coach-led Digital Platform Using an Intelligent Coaching Assistant: A Community Pilot Study
Brief Title: Assessing the Feasibility of a Coach-led Digital Platform
Acronym: Connect5
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Royal College of Surgeons, Ireland (Other)
Responsible Party: Sponsor
Other Study IDs: Connect5 Pilot
Record Dates: First submitted 2023-10-10; First posted 2023-10-23 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Population; Life Style, Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Residents of Athy, Co. Kildare: Anyone who lives, works or plays in Athy and the surrounding 5 Km who is over 18 years is invited to take part.
  Interventions: Behavioral: Human coach-led digital health platform

INTERVENTIONS:
Behavioral: Human coach-led digital health platform — This is an existing commercial digital platform developed by our technology partners (Empeal). The platform comes in the form of a smartphone app available via Android and Apple devices. Participants will communicate with their coach through the app via video, audio or text. Surveys are conducted on the app. Support content is also available through this app.

SUMMARY:
This research is taking place to find out if a smartphone app plus a health coach can support citizens of Athy, Co. Kildare Ireland to make healthy changes in your lifestyle - small changes for better health. This is the first study of its kind in Ireland; Athy is the first town to take part.

Connect5 Athy smartphone app will have a health coach who will advise and support participants make new healthy lifestyle habits linked to sleep, managing stress, increasing physical activity, support healthy eating, cultivate positive local relationships, and help to avoid risky substances like tobacco and alcohol.

This is a 6-month observational study that will be conducted between May and October 2024.

DETAILED DESCRIPTION:
Title: Assessing the feasibility of a coach-led digital platform using an intelligent coaching assistant: A community pilot study.

1. Background The recent global pandemic has highlighted the need for health and wellness interventions that are freely accessible from a person's home; likewise, studies have shown that citizens with lifestyle related diseases are more vulnerable to infections such as COVID-19. The goal therefore is to provide accessible, expert-led motivational support to Irish citizens who need help in the community in relation to promoting healthy lifestyle and preventing lifestyle-related diseases. This pilot study is a continuation of the previously approved 'RCSI Coach Connect project' that examined the impact of a similar online coach-led app on frontline healthcare workers. Lessons from RCSI Coach Connect have shown us that intelligent assistance is required to help human coaches scale this online health solution to larger citizen groups. This project will involve a close collaboration between existing partners: the RCSI Centre for Positive Psychology and Health and Empeal in the development and implementation of a coach-led digital support platform augmented by an Intelligent Coaching Assistant (ICA) for 6-months. This digital health platform is a motivational support unit only and is not intended for use or replacement of medical or therapeutic.

   ICA-augmented coaching has the potential to transform the coaching profession. Having ICA as a partner can facilitate human coaches to improve the quality of their work and has the potential to increase accessibility and availability of coaching through lower costs. The ICA of this digital health platform has been developed to take time-consuming administrative tasks from the human coach so that their time can be maximised for scalability. Administrative tasks that ICA have taken include, on-boarding participants, prompting participants to complete assessments and book coaching session, reporting assessment results, and gathering data for the coach (i.e. short, medium and long-term goals and targets, trackability of goals, along with their readiness to change and feelings of achievability and reality towards goals). All data gathered by the ICA is to be utilised by coaches to augment the one-to-one coaching experience between participants and coaches. Data is the lifeblood of ICA and must be protected and managed. The ICA will only gather data provided by the participants, and this data is completely voluntary. By collaborating with Empeal, the investigators will analyse this real-world data and apply it to the development and validation of an ICA-augmented coaching framework.
2. Project Overview Residents of Athy will have the opportunity to on-board onto the digital health platform for the duration of the project (six months). On the platform, they will have access to educational content (of the 6 vital signs of lifestyle medicine - sleep, physical activity, stress management, healthy eating, relationships, and substance use), a health coach, and data from their wearable devices. Participants can engage in gamification aspects of the application such as contests and challenges aimed to promote engagement and adherence to the lifestyle goals set.

In addition to pilot testing the digital health application in Athy, the researchers will provide in person educational sessions in Athy Library to engage with residents in themes like 'what is health coaching', 'how does digital health work', 'managing your stress', 'healthy eating', 'increasing physical activity', 'improving your sleep', 'minimising substance use', and 'engaging with your community for better health'.

Timelines of research outputs Primary outcome/objectives The aim of this study is to examine the feasibility of running a supporting online health-coach-based digital platform for an urban community, over a 6-month period. The study is conducted with partners from SláinteCare Healthy Communities Kildare, Healthy Ireland, and Empeal (technology provider), with an emphasis on vulnerable populations within the community (perinatal women, lone parents, elderly citizens living alone, citizens with chronic disease, recent migrants and the Irish Traveller community).

Primary outcomes:

1. Assess the feasibility of a coach-led digital health platform in an urban community, using CONSORT guidelines for conducting feasibility/pilot projects. Feasibility will be assessed through recruitment rates, number of logins, engagement, and adherence.
2. To assess the implementation of an intelligent coaching assistant (ICA) designed to support the coach.
3. To assess participants' experience of the coach-led digital platform through qualitative interviews and focus groups.

Secondary outcomes/objectives

1. Identify the needs of vulnerable groups (perinatal women, lone parents, elderly citizens living alone, citizens with chronic disease, recent migrants, and the Irish Traveller community) to inform the adaptation of the digital coaching process to facilitate their engagement in future research.
2. Examine changes in mental health of participants using the Perceived Stress Scale (PSS), wellbeing (PERMA-NHL Profiler), and lifestyle medicine vital signs using the American College of Lifestyle Medicine short form assessment. Changes will be examined using the surveys listed above between time one (during onboarding) and at one-month intervals using the smartphone app.

Deliverables:

1. Ethics, GDPR compliance and sponsorship approval (M1)
2. Participants recruitment (M1)
3. Participant consent and onboarding onto the digital health application (M2)
4. Assessments completed by participants at T1 (M2)
5. Mixed-methods feasibility study of the digital health support platform (M2-7)
6. Assessment completed by participants at T2 (M7)
7. Data transfer from Empeal to RCSI (M8)
8. Qualitative Interviews (M8)
9. Data analysis (M9-11)
10. Feasibility study report (M12)
11. Dissemination of summary data reports to all stakeholders (M12)

Milestones:

1. Ethical and sponsorship approval (M1)
2. Participants recruited and onboarded (M2)
3. Feasibility study complete (M7)
4. Qualitative Interviews complete (M8)
5. Qualitative and quantitative data analysis (M11)
6. Completion and dissemination of feasibility study report (M12)

ELIGIBILITY:
Inclusion Criteria:

* Any citizen who lives works or plays in Athy or the surrounding hinterland and townlands within a 5 KM radius of the town centre
* Over 18 years of age

Exclusion Criteria:

* Not meeting inclusion criteria

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Any citizen who lives works or plays in Athy or the surrounding hinterland and townlands within a 5 KM radius of the town centre. The investigators expect citizens to be of mixed health with some participants having a diagnosis if a noncommunicable chronic disease or other type of chronic diagnosis e.g., heart disease. The remainder are expected to be of general sound health but would like to improve their health status through changes in lifestyle.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Reach of the recruitment process into the target population (community of 9000 citizens). | Month 1
  Reach will be assessed by counting the number of recruited participants as a percentage of the target community, with a population of 9000. This will occur in month 1.
Adoption of the digital platform by study participants during the project | Month 1 to 6
  Adoption will be assessed by calculating the uptake (number of participants who log onto the platform via the smartphone app, compared to those who initially consented), and attrition rates (the number of participants who stopped logging onto the platform via the smartphone app) during the 6 month project.
Engagement as behaviour with the digital health-coaching platform at the end of the 6-month project | Month 1 to 6
  Engagement as behaviour will be assessed by calculating the total login attempts (via the project smartphone app) for each participant at the end of the 6 month project
The experience of a representative number of study participants with the coach-led digital platform, with an emphasis on barriers to and facilitators of engagement using semi-structured interviews | Month 6
  The opinions of a representative number (10%) of study participants will be sought using semi structured interviews (conducted at the end of month 6 with an experienced researcher), using a professional Zoom account. A specific emphasis will be placed on addressing barriers to and facilitators of engagement with the smartphone app and the online coach.

SECONDARY OUTCOMES:
Changes in the perceived stress of participants using the Perceived Stress Scale (PSS). | Month 1 to 6
  Changes in perceived stress of recruits will be examined using the PSS between time one (month 1) and time two (month 6) of the project. Participants will complete this survey at both time points using the dedicated smartphone app.
Changes in wellbeing of participants using the Positive emotion, Engagement, Relationships, Meaning, Accomplishment - Negative emotion, Health, Loneliness (PERMA-NHL) Profiler. | Month 1 to 6
  Changes in the wellbeing of recruits will be examined using the PERMA-NHL Profiler between time one (month 1) and time two (month 6) of the project. Participants will complete this survey at both time points using the dedicated smartphone app.
Changes in healthy lifestyle practices, using the American College of Lifestyle Medicine short form (ACLM-SF) assessment. | Month 1 to 6
  Changes in the healthy lifestyle practices (sleep, eating healthy food, physical activity, stress management, limiting alcohol and tobacco consumption and cultivating positive relationships) of recruits will be examined using the ACLM-SF assessment between time one (month 1) and time two (month 6) of the project. Participants will complete this survey at both time points using the dedicated smartphone app.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal College of Surgeons in Ireland, University of Medicine and Health Sciences, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No
We will publish aggregate summary anonymous data on Zenodo.com.